CLINICAL TRIAL: NCT02548442
Title: Children's Autism Metabolome Project (CAMP): Development and Clinical Evaluation of the Stemina Metabolic Biomarker-Based Test to Diagnose Autism Spectrum Disorder in Early Childhood
Brief Title: Children's Autism Metabolome Project
Acronym: CAMP-01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stemina Biomarker Discovery, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Nancy Lurie Marks Family Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CAMP-01; R44MH107124-01 (NIH)
Record Dates: First submitted 2015-09-02; First posted 2015-09-14 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Autism Spectrum Disorder; Developmental Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma for metabolite analysis and blood samples for DNA and RNA expression analysis will be collected from all children as part of the study protocol. Genetic analysis of samples will be performed only on subjects that have consented to allow this evaluation. In addition, a urine sample for metabolite analysis will also be obtained from children capable of providing the sample while at the clinical site.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Autism Spectrum Disorder: Subjects identified as having Autism Spectrum Disorder using behavioral based methods.
- Developmental Delay: Subjects identified as having a developmental delay that is not Autism Spectrum Disorder using behavioral methods.
- Typically Developing Children: Subjects identified as not having a developmental delay or autism spectrum disorder using behavioral methods as well as not having another serious medical or psychological condition.

SUMMARY:
Development and Clinical Evaluation of the Stemina Metabolic Biomarker-Based Test to Diagnose Autism Spectrum Disorder in Early Childhood.

DETAILED DESCRIPTION:
The purpose of this study is to identify metabolitic signatures in blood plasma and/or urine using a panel of biomarker metabolites that differentiate children with autism spectrum disorder (ASD) from children with delayed development (DD) and/or typical development (TD), to develop an algorithm that maximizes sensitivity and specificity of the biomarker profile, and to evaluate the overall algorithm as a diagnostic tool.

A secondary objective is to define metabolites capable of classifying subtypes of ASD that may increase understanding of the metabolic basis of the condition, as well as inform on personalized therapy.

The population targeted for this study includes children aged 18 months to 48 months, diagnosed with ASD or DD using behavioral criteria, and TD children, identified as having no indications of ASD or DD using behavioral criteria. The original target size for the study was 1500 subjects divided equally between the three groups. The targeted male:female ratio is 4:1 in all three groups. During the study, it was determined that biomarkers capable of identifying ASD subjects could be obtained using a total of 1100 subjects divided with 58% ASD, 25%TD, and 17% DD. If the diagnostic biomarkers identified in the study do not perform well in females during the biomarker discovery phase, the study may be expanded to recruit more females to examine the possibility of a female-specific diagnostic test.

Subjects will be qualified for entry into the study and will be invited to participate. On the first study day, subjects' parents will sign an informed consent form and will be asked questions on the mother's pregnancy and of both parents' medical history. A complete medical history, a physical examination, and information needed to obtain a diagnosis of ASD, DD, or TD will be obtained on the study subject. If possible, a urine sample will be collected during the visit. Up to four tubes of blood (<25 mLs total) will be drawn at the clinic during the visit or within 14 days following this initial visit. An overnight fast is required prior to the visit where blood will be taken from the subject. A subset of the subjects will be asked to return to the clinic 30-60 days later to obtain a replicate metabolic profile.

The study will be divided into a biomarker discovery/method development phase followed by a validation phase of the analytical methods and algorithm that will be used in the clinical test.

The subjects will be randomized and divided equally between a discovery/training set and a validation set. The training set will be used for discovery of the biomarkers and development of the analytical methods intended for the diagnostic test. The validation sample set will be used to evaluate performance of the final clinical methods and algorithms.

Consent will also be sought from all subjects for follow-up contact up to 5 years following enrollment of the last subject enrolled to determine the accuracy of the original behavioral diagnosis over time. Subjects chosen for follow-up will be identified based on the strength of the diagnosis from the behavioral scores and physician assessments as well as the biomarker profiles observed in individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age of greater or equal to 18 months and less than or equal to 48 months
* Fulfills the definition of an autism spectrum disorder, developmentally delayed, or typically developing child in the age range 18-48 months, as determined by a clinician or certified practitioner of the appropriate tests and who is knowledgeable in the field; and
* Has parental (or other legal guardian ) informed consent to participate.

Exclusion Criteria:

* Diagnosis with a chronic condition that could interfere with a diagnosis of ASD or DD, (e.g.: a known history of Fragile X, Rett syndrome, Down syndrome, tuberous sclerosis, trisomy 21, inborn errors of metabolism or other genetic disorder that includes some symptoms of autism)
* Fetal alcohol syndrome, or other serious neurological disorder
* Other serious metabolic disorder, psychiatric disorder, or medical condition involving the liver, kidney, pulmonary, cardiovascular or endocrine systems
* A second child within a family in which a sibling has already been enrolled.
* A child who has previously participated in the CAMP-01 study

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be identified as autism spectrum disorder (ASD) or developmentally delayed (DD) subjects by standard behavioral techniques; Typically developing (TD) subjects will be recruited from the communities in which the autism research centers are situated. The ADOS-2 (research reliable), the Mullen Scales of Early Learning (MSEL), as well as an evaluation based on the DSM-V checklist will be administered to each subject enrolled in the study suspected to have a developmental delay or autism. Typically developing children enrolled in the study will be given an MSEL and a Social Communications Questionnaire (SCQ) evaluation to document that they are neither ASD nor DD subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1102 (Actual)
Dates: Start 2015-08; Primary Completion 2023-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Metabolites in plasma indicative of autism spectrum disorder. | Within 60 months of sample collection
  Study participants were randomized into two independent groups: a biomarker discovery/method development (training set) and a validation set. The validation set is used to assess the performance of the biomarkers identified in the training set once the analytical methods and algorithms are developed using the training set. These biomarkers and algorithms will be used in the clinical diagnostic tests. Using this approach and CLIA validated assays, two diagnostic panels are now able to correctly identify metabolic signatures in 53% of the ASD population in the CAMP study with a specificity of 91% when tested against the validation set of subject samples.

SECONDARY OUTCOMES:
Metabolites in plasma that are specific for subtypes of autism spectrum disorder | Within 60 months of sample collection
  Using the training set or the validation subject set described in the primary aim, the study will seek to identify additional biomarkers such that >75% of the ASD population can be correctly identified with the same high specificity of >90%. In addition, the study will attempt to link the new biomarkers to important metabolic pathways associated with ASD to give insight into the underlying pathophysiologies of the disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Burrier, Ph.D., Principal Investigator — Stemina Biomarker Discovery
Locations (8):
- United States (8):
  - Melmed Center, Scottsdale, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC David MIND Institute, Sacramento, California
  - Lurie Center for Autism, Lexington, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West PR, Amaral DG, Bais P, Smith AM, Egnash LA, Ross ME, Palmer JA, Fontaine BR, Conard KR, Corbett BA, Cezar GG, Donley EL, Burrier RE. Metabolomics as a tool for discovery of biomarkers of autism spectrum disorder in the blood plasma of children. PLoS One. 2014 Nov 7;9(11):e112445. doi: 10.1371/journal.pone.0112445. eCollection 2014. PMID 25380056
- [Result] Smith AM, King JJ, West PR, Ludwig MA, Donley ELR, Burrier RE, Amaral DG. Amino Acid Dysregulation Metabotypes: Potential Biomarkers for Diagnosis and Individualized Treatment for Subtypes of Autism Spectrum Disorder. Biol Psychiatry. 2019 Feb 15;85(4):345-354. doi: 10.1016/j.biopsych.2018.08.016. Epub 2018 Sep 6. PMID 30446206
- [Derived] Smith AM, Donley ELR, Ney DM, Amaral DG, Burrier RE, Natowicz MR. Metabolomic biomarkers in autism: identification of complex dysregulations of cellular bioenergetics. Front Psychiatry. 2023 Oct 2;14:1249578. doi: 10.3389/fpsyt.2023.1249578. eCollection 2023. PMID 37928922